CLINICAL TRIAL: NCT03683771
Title: Assessment of Endometrial Pattern and Sub-endometrial Vascularity in Prediction of Pregnancy Rate in ICSI
Brief Title: Assessment of Endometrial Pattern and Sub-endometrial Vascularity in ICSI Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Other Study IDs: ICSI vascularity
Record Dates: First submitted 2018-09-22; First posted 2018-09-25 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal US with Doppler study — Transvaginal Ultrasound with doppler study on endometrium will be made

SUMMARY:
Despite constant progress in in vitro fertilization (IVF) techniques and ovarian stimulation, pregnancy and embryo implantation rates remain modest . The phenomenon of embryo implantation depends both on the embryo itself and on endometrial receptivity

DETAILED DESCRIPTION:
A favorable uterine medium is necessary for embryo implantation, but endometrial receptivity can be negatively affected by ovarian stimulation . Study of endometrial receptivity is especially limited in the context of IVF cycles .

Biopsy of the endometrium cannot be considered during the treatment, and this has encouraged the development and use of ultrasonography and Doppler-like non-invasive methods to evaluate ovarian response to the stimulation and uterine receptivity .

ELIGIBILITY:
Inclusion Criteria:

- Maternal age from 20 to 40 years. Women with BMI range from 20 - 35 Women diagnosed with primary infertility

Exclusion Criteria:

Maternal chronic medical disorder (diabetes mellitus or hypertension). Women diagnosed with autoimmune diseases or antiphospholipid syndrome

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile women who will undergo ICSI
Study Population: 120 patients will be included in the study whom will meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
The number of patients who will have positive pregnancy rate | within 2 months
  patients who will get pregnant in ICSI cycle with measuring their doppler indices before ovum pick up

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (2):
- Egypt (2):
  - Kasralainy hospital, Cairo
  - Algazeerah and Kasralainy hospital, Giza